CLINICAL TRIAL: NCT01950884
Title: A Randomised Controlled Trial of Lifestyle Versus Ezetimibe Plus Lifestyle in Patients With Non-alcoholic Steatohepatitis
Brief Title: Lifestyle Versus Ezetimibe Plus Lifestyle in Patients With Non-alcoholic Steatohepatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Maurizio R. Averna, MD, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LISTEN; 2013-003465-33 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: •Non-alcoholic Steatohepatitis (NASH)
Keywords: •Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ezetimibe (Experimental): Ezetimibe tablets plus lifestyle
  Interventions: Drug: Ezetimibe; Behavioral: Lifestyle
- lifestyle (Active Comparator): lifestyle
  Interventions: Behavioral: Lifestyle

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe tablets
  Arms: Ezetimibe
Behavioral: Lifestyle — lifestyle

SUMMARY:
* NAFLD (Non-alcoholic fatty liver disease) has become the most common cause of liver disease in Western countries (hepatic manifestation of insulin resistance);
* NAFLD represents a cardiovascular risk factor;
* Lifestyle modification(weight loss)is the effective medical treatment recommended for NASH (Non-alcoholic Steatohepatitis);
* Ezetimibe could represent a novel safe treatment for NAFLD (Patel 2006. Here the investigators propose a Randomized Controlled Pilot Trial to evaluate the addictive effect of ezetimibe on liver histology, biochemical and sonographic parameters in a small (n.40) number of NASH patients randomized for 12 months in two arms: lifestyle vs lifestyle+ezetimibe.

DETAILED DESCRIPTION:
to evaluate the addictive effect of ezetimibe on liver histology, biochemical and sonographic parameters in a small (n.40) number of NASH patients randomized for 12 months in two arms: lifestyle vs lifestyle+ezetimibe.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients older 18 years
* 2.Histological diagnosis of possible or definite NASH, according to Kleiner scorw, within 6 months before randomization -

Exclusion Criteria:

* 1)Average alcohol consumption > 20 g per day in women and > 30 g per day in men
* 2)other causes of chronic liver disease 3) History of or planned gastrointestinal bypass or any additional bariatric surgery/intervention 4)Hepatic cirrhosis with Child-Pugh score of B or C, and/or concomitant HCC 5)Recent(within 6 months) or concomitant use of agents known to cause hepatic steatosis 7)Recent(within 6 months)change in dose/regimen or first treatment with vitamin E, C, betaine, s-adenosylmethionine, ursodeoxycholate, sylimarin, fibrate, statin, pentoxyfilline, angiotensin II inhibitors, orlistat, sibutramine 8)Ongoing or recent therapy (within 6 months) with vitamin D or with medications known to affect vitamin D3 metabolism 9)Any additional condition that might interfere with optimal partecipation in the study, according to Investigators opinion; 10)Be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
HISTOLOGICAL IMPROVEMENT IN THE SEVERITY OF NASH | 52 WEEKS
  1. either improvement in NAS by at least 2 points spread across at least 2 of the NAS components or post-treatment NAS of 3 points or less;
  2. at least 1 point improvement in the score for ballooning degeneration;
  3. no worsening of the fibrosis score.

SECONDARY OUTCOMES:
Changes in individual components of NAS score | 6 weeks, 24 weeks, 52 weeks
  Changes in:
  1. steatosis, lobular inflammation and hepatocellular balloonin;
  2. fibrosis;
  3. serum aminotransferase levels
  4. anthropometric measures, visceral adiposity index (VAI), insulin resistence, lipid profile and liver elastometry.

OTHER OUTCOMES:
Changes in the prevalence and severity of metabolic syndrome and the cardiovascular risk profile (Framingham calculator) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Averna, Professor, Principal Investigator — University of Palermo
Locations (1):
- Dipartimento Biomedico di Medicina Interna e Specialistica Di.Bi.M.I.S., Palermo, Italy, Italy

REFERENCES:
- [Background] Hughes EA, Tracey I, Singhal S, Patel J. Unexpected beneficial effect in the use of ezetimibe in non-alcoholic fatty liver disease. Med Hypotheses. 2006;67(6):1463-4. doi: 10.1016/j.mehy.2006.05.041. Epub 2006 Jul 10. No abstract available. PMID 16831521
- [Background] Petta S, Muratore C, Craxi A. Non-alcoholic fatty liver disease pathogenesis: the present and the future. Dig Liver Dis. 2009 Sep;41(9):615-25. doi: 10.1016/j.dld.2009.01.004. Epub 2009 Feb 14. PMID 19223251
- [Background] Marchesini G, Bugianesi E, Forlani G, Cerrelli F, Lenzi M, Manini R, Natale S, Vanni E, Villanova N, Melchionda N, Rizzetto M. Nonalcoholic fatty liver, steatohepatitis, and the metabolic syndrome. Hepatology. 2003 Apr;37(4):917-23. doi: 10.1053/jhep.2003.50161. PMID 12668987
- [Background] Bedogni G, Miglioli L, Masutti F, Tiribelli C, Marchesini G, Bellentani S. Prevalence of and risk factors for nonalcoholic fatty liver disease: the Dionysos nutrition and liver study. Hepatology. 2005 Jul;42(1):44-52. doi: 10.1002/hep.20734. PMID 15895401
- [Background] Ekstedt M, Franzen LE, Mathiesen UL, Thorelius L, Holmqvist M, Bodemar G, Kechagias S. Long-term follow-up of patients with NAFLD and elevated liver enzymes. Hepatology. 2006 Oct;44(4):865-73. doi: 10.1002/hep.21327. PMID 17006923
- [Background] Fassio E, Alvarez E, Dominguez N, Landeira G, Longo C. Natural history of nonalcoholic steatohepatitis: a longitudinal study of repeat liver biopsies. Hepatology. 2004 Oct;40(4):820-6. doi: 10.1002/hep.20410. PMID 15382171
- [Background] Adams LA, Lymp JF, St Sauver J, Sanderson SO, Lindor KD, Feldstein A, Angulo P. The natural history of nonalcoholic fatty liver disease: a population-based cohort study. Gastroenterology. 2005 Jul;129(1):113-21. doi: 10.1053/j.gastro.2005.04.014. PMID 16012941
- [Background] Targher G, Marra F, Marchesini G. Increased risk of cardiovascular disease in non-alcoholic fatty liver disease: causal effect or epiphenomenon? Diabetologia. 2008 Nov;51(11):1947-53. doi: 10.1007/s00125-008-1135-4. Epub 2008 Sep 2. PMID 18762907
- [Background] Promrat K, Kleiner DE, Niemeier HM, Jackvony E, Kearns M, Wands JR, Fava JL, Wing RR. Randomized controlled trial testing the effects of weight loss on nonalcoholic steatohepatitis. Hepatology. 2010 Jan;51(1):121-9. doi: 10.1002/hep.23276. PMID 19827166
- [Background] Hickman IJ, Jonsson JR, Prins JB, Ash S, Purdie DM, Clouston AD, Powell EE. Modest weight loss and physical activity in overweight patients with chronic liver disease results in sustained improvements in alanine aminotransferase, fasting insulin, and quality of life. Gut. 2004 Mar;53(3):413-9. doi: 10.1136/gut.2003.027581. PMID 14960526
- [Background] Sanyal AJ, Chalasani N, Kowdley KV, McCullough A, Diehl AM, Bass NM, Neuschwander-Tetri BA, Lavine JE, Tonascia J, Unalp A, Van Natta M, Clark J, Brunt EM, Kleiner DE, Hoofnagle JH, Robuck PR; NASH CRN. Pioglitazone, vitamin E, or placebo for nonalcoholic steatohepatitis. N Engl J Med. 2010 May 6;362(18):1675-85. doi: 10.1056/NEJMoa0907929. Epub 2010 Apr 28. PMID 20427778
- [Background] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Background] Musso G, Gambino R, Cassader M, Pagano G. A meta-analysis of randomized trials for the treatment of nonalcoholic fatty liver disease. Hepatology. 2010 Jul;52(1):79-104. doi: 10.1002/hep.23623. PMID 20578268
- [Background] Subramanian S, Goodspeed L, Wang S, Kim J, Zeng L, Ioannou GN, Haigh WG, Yeh MM, Kowdley KV, O'Brien KD, Pennathur S, Chait A. Dietary cholesterol exacerbates hepatic steatosis and inflammation in obese LDL receptor-deficient mice. J Lipid Res. 2011 Sep;52(9):1626-35. doi: 10.1194/jlr.M016246. Epub 2011 Jun 20. PMID 21690266
- [Background] Davies JP, Scott C, Oishi K, Liapis A, Ioannou YA. Inactivation of NPC1L1 causes multiple lipid transport defects and protects against diet-induced hypercholesterolemia. J Biol Chem. 2005 Apr 1;280(13):12710-20. doi: 10.1074/jbc.M409110200. Epub 2005 Jan 25. PMID 15671032
- [Background] Chan DC, Watts GF, Gan SK, Ooi EM, Barrett PH. Effect of ezetimibe on hepatic fat, inflammatory markers, and apolipoprotein B-100 kinetics in insulin-resistant obese subjects on a weight loss diet. Diabetes Care. 2010 May;33(5):1134-9. doi: 10.2337/dc09-1765. Epub 2010 Feb 25. PMID 20185740
- [Derived] Noto D, Petta S, Giammanco A, Spina R, Cabibbi D, Porcasi R, Caldarella R, Ciaccio M, Muratore R, Cefalu AB, Craxi A, Averna M. Lifestyle versus ezetimibe plus lifestyle in patients with biopsy-proven non-alcoholic steatohepatitis (LISTEN): A double-blind randomised placebo-controlled trial. Nutr Metab Cardiovasc Dis. 2022 May;32(5):1288-1291. doi: 10.1016/j.numecd.2022.01.024. Epub 2022 Jan 29. PMID 35256232